CLINICAL TRIAL: NCT06182488
Title: Safety and Efficacy of Enhanced Recovery After Surgery (ERAS) in Patients Undergoing Emergency Laparotomy: A Single Center Randomized Controlled Trial
Brief Title: Enhanced Recovery After Surgery (ERAS) in Patients Undergoing Emergency Laparotomy
Acronym: ERAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Hospital (Other)
Responsible Party: Principal Investigator, Jianing Lu, Director, Tianjin Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-YLS-010; 2023-YLS-010 (Other: Tianjin Hospital)
Record Dates: First submitted 2023-11-21; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Acute Abdomen; Abdominal Trauma; Emergency Surgery
Keywords: Enhanced recovery after surgery (ERAS); Emergency surgery; Acute abdominal disease; Combined anesthesia; Goal-directed fluid therapy
MeSH Terms: conditions — Abdomen, Acute; Abdominal Injuries

STUDY DESIGN:
Intervention Model Description: A single center randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS Group (Experimental): According to the ERAS guidelines, the ERAS group received ERAS protocol.
  Interventions: Other: ERAS protocols
- Conventional group (Other): Conventional perioperative interventions
  Interventions: Other: Conventional protocols

INTERVENTIONS:
Other: ERAS protocols — ERAS protocols for emergency abdominal surgery
  Arms: ERAS Group
Other: Conventional protocols — Conventional protocols for emergency abdominal surgery
  Arms: Conventional group

SUMMARY:
The goal of this clinical trial is to test the safety and effectiveness of the ERAS protocols compared to a conventional care protocols in patients who received emergency laparotomy. The main question it aims to answer are:

• Can the ERAS protocols be used safely and effectively in patients undergoing emergency laparotomy? Participants will be randomised into the ERAS group and the conventional group and will be given the ERAS protocols and the conventional protocols in the perioperative period.

Researchers will compare the ERAS group with the conventional group to see if the ERAS programme is effective.

DETAILED DESCRIPTION:
Since Kehlet first proposed enhanced recovery after surgery (ERAS) protocols in the 1990s, researchers have been widely adopted. Preoperative counseling, standardized anesthesia management protocols, more optimal postoperative analgesic regimens, restriction of intubation and catheterization, early postoperative mobilization, and early oral intake of food are all part of ERAS programs. These programs began in colorectal surgery and have now been expanded to other surgical specialties. Several studies have shown that patients benefit from ERAS programs, including reduced pain, faster return to bowel function, shorter hospital stays, and lower health care costs. However, investigators found that ERAS programs are rarely used for emergency surgery.

Emergency surgery is the treatment of choice for acute abdominal conditions such as traumatic liver rupture, traumatic splenic rupture, and complete bowel obstruction. Nevertheless, investigators found that most clinical studies of ERAS excluded patients who underwent emergency surgery. This is because most researchers probably believe that emergency surgery does not allow enough time for ERAS-related preoperative preparation. In fact, some ERAS programs can be used for emergency surgery, such as the anesthetic modality of combined anesthesia, postoperative multimodal analgesia, earlier postoperative oral feeding and ambulation, and earlier removal of invasive catheters. However, few studies have focused on the use of ERAS in emergency surgery.

The present study is a randomized controlled trial evaluating the safety and efficacy of an ERAS program in emergency abdominal surgery. Investigators hypothesized that an ERAS program could be implemented into emergency surgery and reduce postoperative recovery time without increasing the complication rate and readmission rate (<30 days).

The standard operating procedures for the study are as follows:

* Participants will be randomised into the ERAS group and the conventional group.
* Preoperative care: A number of preoperative protocols were similar in both groups, including (1) surgical risk assessment; (2) preoperative placement of a nasogastric tube (NG); (3) preoperative administration of crystalloid fluids to replenish blood volume; (4) empiric antibiotics and acid-reducing therapy administered intravenously; and (5) intravenous analgesia.

In the ERAS group, an epidural catheter was placed in the lumbar 3-4 space before surgery to facilitate intraoperative epidural anaesthesia and postoperative analgesia. At the same time, ultrasound-guided internal jugular vein (IJV) cannulation was performed to monitor central venous pressure (CVP). CVP-guided infusion, i.e., goal-directed fluid therapy, was maintained at a CVP of 8-10 cm of saline. Depending on the urinary output, blood pressure, heart rate, and clinical signs of dehydration, fluids were administered according to an institutional care plan in the routine care group. Dexamethasone 4 mg IV was given shortly before induction of anaesthesia.

* Intraoperative care: All patients underwent emergency open surgery. Appropriate surgical incisions were selected based on adequate provision of good surgical vision and surgical space. If intra-abdominal fluid was found, it was aspirated and sent for bacterial culture. The final decision on the surgical approach is based on the surgeon's opinion and intraoperative findings. If anastomosis was deemed unsafe, an ileostomy without anastomosis was performed. Table 1 shows the changes in the anaesthesia regimen in the ERAS group. The anesthesiologist decided on the anaesthesia for the conventional group. In the ERAS group, an experienced surgeon set up an abdominal drain as needed during the procedure. In the conventional care group, an abdominal drain was routinely placed.
* Postoperative care: Patients in the ERAS group were asked to start simple bed activities, such as moving both lower limbs, on the day of surgery (POD-0), provided that the epidural catheter was secure. At POD-1, patients were asked to sit for at least 2 hours and then get out of bed after the epidural catheter was removed at POD-2. In the conventional group, patients were encouraged to be active at POD-2, starting with simple bed activities and gradually transitioning to normal walking without any specific requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages 18-70,
* Patients who completed the preoperative examination and preoperative diagnosis within 4 hours after admission for acute abdomen diseases,
* Required emergency surgery within 6 hours from surgeon encounter.

Exclusion Criteria:

* Patients who refused to be enrolled in this study;
* Patients with any psychiatric or neurological disorders;
* Pseptic shock at admission;
* Duration of symptoms more than five days;
* Patients with contraindications to the placement of lumbar epidural catheters, such as coagulation disorders, severe sepsis, etc.;
* Presence of preoperative factors affecting wound healing (e.g. long-term steroid use);
* Patients with extra-abdominal injuries or terminal malignancy, or patients requiring damage control surgery;
* Patients found intraoperatively to require any procedure other than splenectomy, partial hepatectomy or liver repair, bowel resection and anastomosis, laparoscopic cholecystectomy and appendectomy, and gastrointestinal perforation repair.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
postoperative recovery time | From enrollment to the end of treatment at 2 weeks
  Postoperative recovery time that meets the relevant definitions in this study

SECONDARY OUTCOMES:
the rate of postoperative complications | From enrollment to the end of treatment at 2 weeks
  Percentage of participants who met the recovery condition after surgery as a percentage of total participants
The time of first postoperative flatus | From enrollment to the end of treatment at 2 weeks
  The time of first postoperative flatus
The time to tolerate semi-fluid diet after surgery | From enrollment to the end of treatment at 2 weeks
  The time to tolerate semi-fluid diet after surgery
The time to tolerate soft food after surgery | From enrollment to the end of treatment at 2 weeks
  The time to tolerate soft food after surgery
The rate of readmission (in 30 days) | From enrollment to the end of treatment at 2 weeks
  Percentage of participants who were readmitted to the hospital within 30 days after surgery for an adverse event related to this procedure as a percentage of total participants

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zheng, MD, Study Chair — Tianjin First Central Hospital
Locations (1):
- Tianjin Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT06182488/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT06182488/ICF_001.pdf